CLINICAL TRIAL: NCT05120544
Title: Expanding Technology-Enabled Nurse Delivered Chronic Disease Care
Acronym: EXTEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRO00107722; 1R01NR019594-01 (NIH)
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization will occur following the baseline appointment. We will not blind participants to arm assignment because they will receive information on both arms during consent. In order to assure blinding of staff conducting outcome data collection, randomization will be managed by staff members not involved with outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXTEND (Active Comparator): EXTEND participants receive 4 mobile monitoring devices to facilitate chronic disease self-management (glucometer, BP cuff, scale, accelerometer). Device data are transferred to Duke University Health System (DUHS). Participants can review data and trends within the device apps and modify self-management practices accordingly. The EXTEND group continues chronic disease care with their existing providers during the study, and are instructed at baseline to address management questions via their primary clinics' established avenues (as would be the case for any patient using mobile monitoring in clinical practice).
  Interventions: Behavioral: EXTEND
- EXTEND Plus (Experimental): EXTEND Plus participants receive 4 mobile monitoring devices to facilitate chronic disease self-management (glucometer, BP cuff, scale, accelerometer). Device data are transferred to Duke University Health System (DUHS) for use as part of nurse-delivered intervention combining mobile monitoring, self-management support, and medication management. The intervention is administered by clinical registered nurses (RNs) from Duke Primary Care (DPC) or Duke Endocrinology. For the medication management component, RNs work with a study PharmD affiliated with the participant's clinic. The PharmD determines if medication changes are needed, and prescribes accordingly. The RNs deliver EXTEND Plus via scheduled telephone encounters throughout the 12-month intervention. The initial encounter frequency is every two weeks, but may be extended to every four weeks for patients achieving treatment goals.
  Interventions: Behavioral: EXTEND Plus

INTERVENTIONS:
Behavioral: EXTEND Plus — The EXTEND Plus approach builds patient self-management capacity by focusing on knowledge, self-efficacy, and goal setting (using an RN-delivered, module-based approach). All material is at an 8th grade reading level. Module topics include, but are not limited to, use of self-monitoring of blood glucose (SMBG), BP monitoring, developing a diet plan, medication adherence, hypoglycemia and hypotension self-management, and self-managing insulin. In addition, this intervention component addresses diet and activity self-management during each encounter.
  Arms: EXTEND Plus
Behavioral: EXTEND — EXTEND patients self-manage using data they collect during the study, and continue to receive standard behavioral counseling from primary providers.
  Arms: EXTEND

SUMMARY:
The purpose of this study is to investigate whether the self-management of diabetes and hypertension can be improved with the use of mobile monitoring devices and nursing support.

DETAILED DESCRIPTION:
EXpanding Technology-Enabled, Nurse-Delivered Chronic Disease Care (EXTEND) seeks to address evidence gaps that prevent practical use of mobile monitoring-enabled telehealth for clinic-refractory chronic diseases, with an initial focus on Persistent Poorly Controlled Diabetes Mellitus (PPDM) and hypertension. Because our population has already proven refractory to usual care, we will conduct an active comparator randomized trial (N=220) of two 12-month interventions: 1) mobile monitoring as a self-management tool (EXTEND); and 2) a nurse-delivered intervention incorporating mobile monitoring, self-management support, and medication management (EXTEND Plus). The medication management is a care team approach where the nurse works with a Pharmacist who has prescribing rights to optimize medications for the patients. This proposal will also allow us to examine a novel application for mobile monitoring technologies, as tools for predicting patient safety events.

Aim 1: Compare the effectiveness of the two 12-month EXTEND interventions for PPDM and hypertension. Hypothesis 1a: Compared to EXTEND, EXTEND Plus will improve primary (HbA1c) and secondary outcomes (e.g., blood pressure, weight, self-management measures) at 12 months; Hypothesis 1b: The relative effects of each intervention will be sustained at 24 months; Hypothesis 1c: Subgroup analyses will identify characteristics associated with high responsiveness to each intervention.

Aim 2: Guide scaling and dissemination of the EXTEND interventions by: (A) interviewing patients and stakeholders to clarify implementation barriers, facilitators and process requirements; (B) comparing intervention costs against potential reimbursement mechanisms; and (C) understanding the role of climate change and other social drivers of health on diabetes self-management and intervention engagement.

Aim 3: Explore the value of combining mobile monitoring and EHR data for predicting patient safety events (hospitalizations, emergency visits) in the EXTEND study cohort over 24 months. Participants will monitor their data using a suite of remote monitoring devices. Data will be analyzed with PACE by our team. If participants are randomized to the telehealth arm, these data will be reviewed by a RN during a telehealth visit to aid in clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes by International Classification of Diseases (ICD) code or treatment with glucose-lowering medication or mention in clinical notes
* Poor diabetes control as indicated by at least 1 HbA1c greater than or equal to 8.0% with NO HbA1c less than 8.0% over the past 6 months
* At least 1 appointment (office visit, appointment, initial consult, telemedicine) at primary clinic site over the past year
* hypertension by ICD code or treatment with blood pressure-lowering medication or mention in clinical notes
* poor hypertension control as indicated by a clinic systolic BP >140 AND/OR diastolic BP >90 over past year
* use of an Apple iPhone or Android smartphone
* can provide informed consent
* can read/speak English
* can provide informed consent

Exclusion Criteria:

* dementia, psychosis, or life-limiting illness
* acute coronary event in past year
* hypoglycemic seizure/coma over the past year
* residence in a nursing home
* use of an insulin pump
* are or plan to become pregnant
* unable or unwilling to use necessary technology to participate in study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline, 3, 6, 9, 12, 18 and 24 months
  Change in blood sugar (glucose) attached to hemoglobin. Validated point-of-care or lab-based test.

SECONDARY OUTCOMES:
Change in blood pressure | Baseline, 3, 6, 9, 12, 18 and 24 months
  Measure taken at clinic with standard arm cuff. Measurement is the average of two readings, on the same arm, taken 10 minutes apart.
Change in weight | Baseline, 3, 6, 9, 12, 18 and 24 months
  Measurement taken with lab scale, when patient is lightly clothed, shoes off.
Change is Diabetes Distress Scale | Baseline, 6, 12, 18 and 24 months
  Measure of diabetes distress and burden using the Diabetes Distress Scale (DDS): 17 items, Scale 1-6. Scoring: Average. Higher score indicates higher distress level.
Change in Diabetes Self-Management Questionnaire | Baseline, 6, 12, 18 and 24 months
  Measure of diabetes self-care. Diabetes Self-Management Questionnaire (DSMQ): 16 items, Scale 0-3. Scoring: Sum and transform to fall between 0-10. Higher score indicates more effective self-care.
Change in Perceived Competence Scale | Baseline, 6, 12, 18 and 24 months
  Measure of diabetes self-efficacy and capacity. Perceived Competence Scale (PCS): 4 items, Scale 1-7. Scoring: average (1-7) Higher score indicates greater self-efficacy.
Change in medication non-adherence | Baseline, 6, 12, 18 and 24 months
  Validated self-report measure using Voils' medication non-adherence measure.
Change in diabetes knowledge | Baseline, 6, 12, 18 and 24 months
  Diabetes Knowledge Questionnaire (DKQ) is a 24-item validated measure.
Change in hypertension knowledge | Baseline, 6, 12, 18 and 24 months
  Hypertension Knowledge Measure (HKM) is an 11-item validated measure.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Shaw, RN, PhD, Principal Investigator — Duke University School of Nursing; Matthew Crowley, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Our data will be made available for use by investigators not associated with the proposed study within 3 years after the primary results have been published. We will prepare a clear and searchable documentation of the database including a data dictionary, and its linkage to the pertinent study protocols and forms so that diverse investigators can make effective use of the data. For investigators interested in prospective collaborations, we will explore other options to provide support.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Within 3 years of study data publication.
Access Criteria: For all prospective opportunities (e.g., access to datasets, collaborative studies), we will widely advertise them on Duke Websites and at appropriate scientific meetings.

REFERENCES:
- [Derived] Lee D, Yang Q, Crowley MJ, Hatch D, Pennington G, Matters D, Shaw RJ. Chronic Illness Self-Management Latent Profiles in Individuals With Comorbid Type 2 Diabetes and Hypertension. Sci Diabetes Self Manag Care. 2025 Jun;51(3):250-261. doi: 10.1177/26350106251336311. Epub 2025 May 14. PMID 40370006

DOCUMENTS (1):
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT05120544/ICF_000.pdf